CLINICAL TRIAL: NCT04724993
Title: Comparison the Effectiveness of Online Aerobic Dance Exercises Versus Physical Activity Counseling in Patients With Juvenile Familial Mediterranean Fever
Brief Title: Effects of Online Aerobic Exercise Training and Physical Activity Counseling in Juvenile Familial Mediterranean Fever
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Istanbul University (Other)
Responsible Party: Principal Investigator, Saime Nilay Arman, Assist.Prof., Istanbul University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 05/12/2019-186585
Record Dates: First submitted 2021-01-22; First posted 2021-01-26 (Actual); Last update posted 2021-01-26 (Actual); Status verified 2021-01

CONDITIONS: Familial Mediterranean Fever; Exercise; Physical Activity
Keywords: Familial Mediterranean Fever; Online Exercise; Physical Activity Counseling; Aerobic Dance
MeSH Terms: conditions — Familial Mediterranean Fever; Motor Activity

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Online Aerobic Dance Exercises (Experimental): In this group, aerobic dance exercises will be applied online under the supervision of a physiotherapist. And participants will record their physical activities on the Physical Activity Tracking Chart.
  Interventions: Other: Online Aerobic Dance Exercises
- Physical Activity Counseling (Experimental): In this group, participants will be informed online about physical activity and exercise. And they will record their physical activities on the Physical Activity Tracking Chart too.
  Interventions: Other: Physical Activity Counseling

INTERVENTIONS:
Other: Online Aerobic Dance Exercises — Online aerobic dance exercises will be performed with observance of physiotherapist. They will record their daily physical activity.
  Arms: Online Aerobic Dance Exercises
Other: Physical Activity Counseling — Physical activity and exercise will ve explained to the participants.And they will record their daily physical activity.
  Arms: Physical Activity Counseling

SUMMARY:
The aim of the study is to investigate comparison the effectiveness of online aerobic dance exercises versus physical activity counselling in patients with Juvenile Familial Mediterranean Fever.

ELIGIBILITY:
Inclusion Criteria:

* To be under colchicine treatment for at least 3 months
* Being in an attack-free period

Exclusion Criteria:

* Attack in the last 2 weeks
* Having any systemic chronic disease except Familial Mediterranean Fever
* Presence of amyloidosis
* Having arthritis that may prevent participation in exercise

Ages: 8 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 30 (Actual)
Dates: Start 2020-12-20 (Actual); Primary Completion 2021-02 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Six Minute Walk Test | Change from baseline to 8 weeks
  The 6-minute walk test is a well tolerated, easy-to-apply and a simple test that shows the submaximal level of functional capacity. This test measures the distance that patients can walk quickly on a hard and flat surface within 6 minutes. Patients will be rested in a chair near by the starting position for at least 10 minutes before the test begins. Heart rate, blood plessure, saturation and fatigue levels will be determined by a physiotherapist before and after the test. At the end of the test, the distance walked by the patients within 6 minutes will be recorded in meters.

SECONDARY OUTCOMES:
Progressive Aerobic Cardiovascular Endurance Run (PACER) | Change from baseline to 8 weeks
  PACER is an adaptation of the 20-meter shuttle running test and it is a field test consisting of multiple stages. Participants will run forward and backward in an area of 20 meters, accompanied by music from a tape recorder. The test will start at slow speeds and the speed will gradually increase every minute. The test will be ended when participants cannot continue to run at the level they have reached. The number of laps completed as a result of the test will be recorded.
Skinfold Thickness Measurement and Bioelectrical Impedance Analysis | Change from baseline to 8 weeks
  FitnessGram uses the triceps and calf areas to measure skinfold thickness, as it is easy to measure and is not too invasive. Measurements will be made with a caliper. And participants' body composition will be evaluated with the Tanita Body Analyzer.
Curl Up Test | Change from baseline to 8 weeks
  Abdominal muscle strength and endurance will be evaluated with curl up test. The goal of this test is to do many curl-ups at a specific rhythm as possible. Maximum 75 curl-ups will be counted. At the end of the test, the number of curl-ups will be recorded.
Trunk Lift Test | Change from baseline to 8 weeks
  Trunk extensor muscle strength and flexibility will be evaluated with trunk lift test. Participants will start the test in the prone position. A mark will be placed on the floor at the participants' eye level. During the test, participants raise their torsos slowly and in a controlled manner to a maximum height of 12 inches. At the end of the test, the distance between the floor and the jaws of the participants will be measured and the score will be recorded in cm.
Push Up Test | Change from baseline to 8 weeks
  Upper extremity muscle strength and endurance will be evaluated with push up test.During the test, participants move their torsos towards the ground, when their elbows are bent at 90º, they raise themselves again. The movement is repeated as much as possible. The rhythm is set to 20 push-ups per minute or 1 push-up per 3 seconds. The number of push-ups performed at the end of the test will be recorded.
Back saver Sit and Reach Test | Change from baseline to 8 weeks
  Hamstring muscles' flexibility will be evaluated with back saver sit and reach test. A box is needed for the test. This box is 35 cm long, 45 cm wide, 32 cm high. A 55 cm long and 45 cm wide top plate is placed on the box. One leg of the participants' is completely straight while the other is bent at the knee. Participants reach forward four times by placing their hands on top of each other, holding the fourth access position for 1 second. The distance will be recorded at the end of the test.
Physical Activity Questionnaire for Older Children (PAQ-C) | Change from baseline to 8 weeks
  This scale, developed by Kowalski et al. in 1997, is a 9-item seven-day recall measurement tool designed to evaluate the general physical activity levels of children and adolescents throughout the school year.
Physical Activity Questionnaire for Adolescents (PAQ-A) | Change from baseline to 8 weeks
  This scale, developed by Kowalski et al. in 1997, evaluates the general physical activity level of high school students aged 14-19. It is a measurement tool consisting of 8 items and based on remembering for seven days.
PedsQL™ Multidimensional Fatigue Scale | Change from baseline to 8 weeks
  The PedsQL Multidimensional Fatigue Scale is an 18-question scale developed to assess fatigue in pediatric patients. It evaluates general fatigue, fatigue during sleep/rest, and cognitive fatigue.
Familial Mediterranean Fever Quality of Life Scale (FMF-QoL) | Change from baseline to 8 weeks
  This scale, developed by Ulutatar and Duruoz, is specific to Familial Mediterranean Fever patients and consists of 20 questions that evaluate the quality of life.
Visual Analogue Scale for Fatigue | Change from baseline to 8 weeks
  A 100 mm VAS will be used to evaluate the fatigue of the participants. Scores <20 mm according to VAS mean "low fatigue", scores between 20-49 mm mean "clinically significant fatigue" and scores with ≥50 mm mean "severe fatigue".
Visual Analogue Scale | Change from baseline to 8 weeks
  It will be used to assess the pain levels of the participants. It is applied by marking with a pencil on a 100 mm horizontal or vertical line. There is no pain at the 0 mm point of this line, and the most severe pain at the 100 mm point.

CONTACTS AND LOCATIONS:
Overall Officials: Saime Nilay ARMAN, Study Director — Istanbul University - Cerrahpasa
Locations (1):
- Istanbul University-Cerrahpasa, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No